CLINICAL TRIAL: NCT04598750
Title: The Neonatal Hemorrhagic Risk Assessment in Thrombocytopenia Study-2
Brief Title: The Neonatal Hemorrhagic Risk Assessment in Thrombocytopenia
Acronym: NEOHAT-2
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Boston Children's Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); Region Stockholm (Other Government); The Swedish Society of Medicine (Other)
Responsible Party: Principal Investigator, Emoke Deschmann, Principal Investigator, Karolinska Institutet
Other Study IDs: TRF15483; 2P01HL046925-21A1 (NIH)
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Neonatal Thrombocytopenia; Bleeding
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study designed to evaluate Immature Platelet Fraction or Immature Platelet Count and Platelet Function Analyzer-100/200 Closure Time-ADP (in vitro bleeding time) as markers of bleeding risk in thrombocytopenic preterm neonates admitted to the Neonatal Intensive Care Unit.

DETAILED DESCRIPTION:
Thrombocytopenia is a known risk factor for clinically significant bleeding in neonates. However, there is a poor correlation between degree of thrombocytopenia and bleeding risk. A better marker of bleeding risk suitable for use in neonates could help physicians more accurately determine the risk/benefit ratio of platelet transfusions, guiding platelet transfusion decisions, and potentially protecting vulnerable infants from exposure to unnecessary transfusion-related risks. The investigators recently found that the Platelet Function Analyzer (PFA) Closure Time-Collagen/ADP (CT-ADP) was a better marker of bleeding than the platelet count in preterm neonates. However, the CT-ADP requires 0.8 mL blood limiting its potential widespread use. The Immature Platelet Fraction (IPF) is a new laboratory marker measuring the % newly released and more active platelets, measured from the same sample as the platelet count. This is a prospective observational study designed to evaluate IPF as marker of bleeding risk in thrombocytopenic neonates admitted to the Neonatal Intensive Care Unit, compared to platelet counts alone. And also, to validate the previously found association between PFA-100/200 CT-ADP and bleeding in a bigger cohort, to compare the IPF with the PFA-100/200 CT-ADP as bleeding predictors and to assess whether the PFA-100/200 CT-ADP combined with the IPF is able to predict bleeding in thrombocytopenic preterm neonates.

ELIGIBILITY:
Inclusion Criteria:

* Have a gestational age <32 weeks and a birth weight ≥500 grams;
* Have a platelet count <100 x 109/L; and
* Have a parent/guardian willing to provide written informed consent.

Exclusion Criteria:

* Are not expected to survive for >24 hours by the Attending Neonatologist;
* Are thought to have a familial thrombocytopenia or platelet dysfunction, based on family history or clinical presentation (associated congenital malformations, platelet morphology).

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Infants will be eligible for study if they have a gestational age <32 weeks and a birth weight ≥500 grams; and have a platelet count <100 x 109/L.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
NeoBAT score | 24 hours
  NeoBAT scores will include any bleeding since the last platelet count or over the prior 24 hours, whichever is shortest. This will serve to correlate bleeding scores (NeoBAT) with platelet counts, IPF% and IPC, PFA-100/200 CT-ADP, and to quantify changes in response to platelet transfusions. The scale is 1 to 4 with 1 being Minor Hemorrhage and 4 being Severe Hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Emöke Deschmann, MD, PhD, Principal Investigator — Karolinska Institutet; Robert Christensen, MD, Study Chair — University of Utah Medical Center
Locations (8):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Intermountain Medical Center, Murray, Utah
  - Utah Valley Hospital, Provo, Utah
- Netherlands (2):
  - Amsterdam University Medical Centre, Amsterdam
  - Leiden University Medical Center, Leiden
- Sweden (2):
  - Karolinska University Hospital Huddinge campus, Huddinge
  - Karolinska University Hospital Solna campus, Astrid Lindgren Children's Hospital, Stockholm